CLINICAL TRIAL: NCT06851065
Title: Luspatercept Treatment Patterns and Outcomes Among ESA-Naïve Patients With Lower-Risk MDS - A Retrospective Medical Record Review in the United States
Brief Title: A Study to Evaluate Luspatercept Treatment Patterns and Outcomes in Erythropoiesis-Stimulating Agents-Naïve Patients With Lower-Risk Myelodysplastic Syndromes in the United States
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA056-1121
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Myelodysplastic Syndromes
Keywords: Lower-risk myelodysplastic syndromes (LR-MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — luspatercept; Hematinics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Participants receiving first-line luspatercept treatment
  Interventions: Drug: Luspatercept
- Participants receiving first-line erythropoiesis-stimulating agents
  Interventions: Drug: Erythropoiesis-stimulating agents

INTERVENTIONS:
Drug: Luspatercept — As per product lable
  Groups: Participants receiving first-line luspatercept treatment
Drug: Erythropoiesis-stimulating agents — As per product label
  Groups: Participants receiving first-line erythropoiesis-stimulating agents

SUMMARY:
The purpose of this study is to understand real-world effectiveness of luspatercept treatment among erythropoiesis-stimulating agents -naïve patients with lower-risk- myelodysplastic syndromes in the United States

ELIGIBILITY:
Inclusion Criteria:

* Had a documented diagnosis of primary or secondary myelodysplastic syndromes (MDS)
* MDS diagnosis confirmed through bone marrow testing on (or 30 days prior to) MDS diagnosis date or within 1 year of MDS diagnosis date
* Had a documented determination of Lower Risk (LR)-MDS as measured by International Prognostic Scoring System (IPSS) or its revised version (IPSS-R) at or before index treatment (i.e., first-line luspatercept or first-line erythropoiesis-stimulating agents (ESA)) initiation

  * IPSS risk level: low, intermediate-1 (level-1 risk)
  * IPSS-R risk level: very low, low, intermediate
* Received luspatercept as the first-line treatment for anemia any time from 28 August 2023 to 31 July 2024 (Cohort 1)

  * Receipt of combination therapy with ESAs and/or granulocyte colony-stimulating factors (G-CSFs) will be allowed

OR

* Received ESA as the first-line treatment for anemia any time from 28 August 2023 to 31 July 2024 (Cohort 2)
* Was aged 18 years or older at the time of initial diagnosis of MDS
* Known vital status (i.e., living, or deceased) at the time of record abstraction.

  * Records for patients who are dead or alive will be eligible
* Complete medical record covering relevant past medical history, diagnosis of LR-MDS, treatment, laboratory assessments, red-blood cell (RBC) transfusions, and regular monitoring for LR-MDS, including any transfer record from other physicians/facilities (if applicable) is available to the abstracting physician for data abstraction

Exclusion Criteria:

* Had a history of acute myeloid leukemia (AML) prior to MDS diagnosis
* Received previous treatment with hypomethylating agents, disease-modifying agents (including lenalidomide), other immunosuppressants/immunomodulatory agents, or other MDS-directed chemotherapy
* Received stem cell transplant prior to index treatment initiation
* Participated in a clinical trial for the treatment of MDS before or while on index treatment (i.e., clinical trial participation after first-line luspatercept or ESA treatment discontinuation will be allowed)
* Had evidence of other malignant neoplasms in the 12 months prior to diagnosis of MDS, except basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, or incidental histologic finding of prostate cancer (stage T1a or T1b)

  * Patients for whom this information is not available (i.e., "unknown") will be included in the study
* For Cohort 1 (i.e., first-line luspatercept treatment), receipt of combination therapy with hypomethylating agents, lenalidomide, other immunosuppressants/ immunomodulatory agents, or other MDS-directed chemotherapy
* For Cohort 2 (i.e., first-line ESA treatment), receipt of combination therapy with hypomethylating agents, lenalidomide, luspatercept, other immunosuppressants/ immunomodulatory agents, or other MDS-directed chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults in the United States with a clinician-confirmed diagnosis of primary or secondary lower-risk myelodysplastic syndromes (LR-MDS) who initiated first-line luspatercept treatment on or after LR-MDS diagnosis date between 28 August 2023 to 31 July 2024
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Participant baseline demographics | Baseline
Participant baseline clinical characteristics | Baseline
Time from Lower Risk- myelodysplastic syndromes diagnosis to index treatment initiation | Baseline
Rationale for therapy selection | Baseline
Duration of index treatment | Up to 15 months
Treatment dose at treatment initiation and discontinuation | Up to 6 months
Treatment dose/dosing schedule changes, and treatment interruptions | Up to 12 months
Other supportive care therapies prescribed while on index treatment | Up to 15 months
Treatments prescribed post index treatment | Up to 15 months
Treatments for anemia management received after discontinuing the index treatment | Up to 15 months
Receipt of stem cell transplant at any time post index treatment | Up to 15 months
Participant red-blood cell (RBC) transfusion burden post index treatment | At 3-months, and up to 6 months
Hematologic improvement-erythroid (HI-E) response post index treatment | At 3-months, and up to 6 months
Progression to acute myeloid leukemia post index treatment | Up to 15 months
Progression to high-risk myelodysplastic syndromes per the International Prognostic Scoring System (IPSS) or its revised version (IPSS-R) criteria | Up to 15 months
Participant adverse events during and post index treatment | Up to 15 months
Overall survival (OS) | At 3-, 6-, 12-, and up to 15-months
Healthcare resource utilization (HCRU) during index treatment | Up to 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- RTI Health Solutions, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts